CLINICAL TRIAL: NCT04341636
Title: A Comparison of the Accurate Diagnosis of the Horizontal & Vertical Bitewing Images in Detecting Approximal Caries and Interdental Bone Loss in Posterior Teeth: A Randomized Controlled Clinical Trial
Brief Title: A Comparison of the Accurate Diagnosis of the Horizontal & Vertical Bitewing Images
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Zuhair Saleh Natto, Head of research unit and assistant professor, King Abdulaziz University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0530517
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Periodontal Diseases; Dental Caries
Keywords: Radiography, Bitewing
MeSH Terms: conditions — Periodontal Diseases; Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vertical bitewing (Experimental): All of the bitewing radiographs will be evaluated by two experienced restorative dentists for caries. All observers will be instructed on the definition of the rating scale before the examination sessions. The observers will be using the following a 5-point confidence scale as follows: 1=caries definitely absent; 2=caries probably absent; 3=equal chance of caries being present or absent; 4=caries probably present; 5=caries definitely present. If caries was detected a second 5-point confidence scale as follows: 1=caries mostly absent (< 25%); 2=caries slightly presence( 25%-50%) ; 3=about half of the border are presence; 4=caries probably clear ( most boarders are presence); 5=caries definitely clear ( all borders are presence ).
  Interventions: Radiation: Bitewing X ray
- horizontal bitewing (Active Comparator): All of the bitewing radiographs will be evaluated by two experienced periodontist for bone loss measurements. The steel wire will be used to determine the magnification factor as explained by G Li et al. 8 The steel wire and cemento enamel junction (CEJ) - if not obscure by caries - will be used as reference points for bone loss measurements. Each tooth will be measured mesially and distally twice and all these measurements will be adjusted using the steel measurement.9 All the measurements will be conducted using IC measure INK software.
  Interventions: Radiation: Bitewing X ray

INTERVENTIONS:
Radiation: Bitewing X ray — Each patients will be exposed to 4 horizontal bitewing for posterior teeth ( standard of care ) and 4 vertical bitewing for the same area ( experimental ) . X ray will be taken using a film holder and a steel wire (3mm ) on the film holders. This steel wire will help to adjust for magnification later on. The x ray tube will be in the same distance (4mm from the x ray).
  The bitewing radiographs will be taken with double-packed Ekta speed Plus films on a radiograph machine operating at 0 kilovolt peak and 8 milliampere, having 2.5 aluminium filtration and a 0.860.8 mm focal spot, according to the manufacturer's exposure recommendations, with the parallel technique to obtain an accurate x ray as much as possible . The radiographs will be processed digitally. All the x ray will be taken using the standard protection protocol .

SUMMARY:
The aims of this research are to determine if vertical bitewings will be more effective and more comprehensive for the diagnosis of caries and the level of alveolar bone loss than the horizontal bitewing technique for the patients at King Abdulaziz University over the age of 18. This is a cross sectional study. All the images in this study will be conducted at School of Dentistry, King Abdulaziz University. Each patients will be exposed to 4 horizontal bitewing for posterior teeth ( standard of care ) and 4 vertical bitewing for the same area ( experimental ). The radiographs will be processed digitally. All the x ray will be taken using the standard protection protocol.

DETAILED DESCRIPTION:
The aims of this research are to determine if vertical bitewings will be more effective and more comprehensive for the diagnosis of caries and the level of alveolar bone loss than the horizontal bitewing technique for the patients at King Abdulaziz University over the age of 18. This is a cross sectional study. All the images in this study will be conducted at School of Dentistry, King Abdulaziz University. Each patients will be exposed to 4 horizontal bitewing for posterior teeth ( standard of care ) and 4 vertical bitewing for the same area ( experimental ) . X ray will be taken using a film holder and a steel wire (3mm ) on the film holders. This steel wire will help to adjust for magnification later on. The x ray tube will be in the same distance (4mm from the x ray). The bitewing radiographs will be taken with double-packed Ekta speed Plus films on a radiograph machine operating at 70 kilovolt peak and 8 milliampere, having 2.5 aluminium filtration and a 0.860.8 mm focal spot, according to the manufacturer's exposure recommendations, with the parallel technique to obtain an accurate x ray as much as possible . The radiographs will be processed digitally. All the x ray will be taken using the standard protection protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age.
2. Patients who are currently be treated KAU dental clinics and meet all medical and dental requirements of the KAU clinic for treatments (e.g., subjects with no diseases contraindicating their dental treatment at KAU).
3. Display no evidence of acute periodontal infection: e.g., abscess, suppuration, severe swelling and/or spontaneous bleeding that required urgent treatment
4. Non-smoker.
5. Patients who have opposing teeth and no missing posterior or canine teeth in all quadrants (except third molars).

Exclusion Criteria:

1. Have any known disease and would not allow the patient to be treatment planned for any procedures in the KAU clinics (e.g., severe anemia, low white blood cell count (Absolute Neutrophil Count (ANC) less than 1500, bleeding or coagulation disorder, uncontrolled hypertension (150/90), recent myocardial infarction (within 6 months of enrollment), diabetes (HbA1C ≥7%), HIV/AIDS (self-reported), history of or currently undergoing head and neck radiation, history of or currently taking bisphosphonates, endocrine-induced bone diseases (e.g. hyperparathyroidism), immunosuppressive therapy).
2. Have limited mental capacity and unable to give informed consent.
3. Be a pregnant or lactating female (self-reported)
4. Have untreated malignant neoplasm.
5. Individuals opposed to participate in the study.
6. If a patient has a crown which will not be able to assess the caries boarder and cementoenamel junction.
7. if a patient has a gagging reflex or inability to open his/her mouth.

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University , Faculty of Dentistry, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 patients were screened for eligibility at the dental clinic
Pre-assignment Details: 20 participants were randomized.
Groups:
- Vertical Bitewing, Then Horizontal Bitewing: Participants first received vertical bitewing in one day for 15 minutes . After a washout period of 10 minutes, they then received horizontal bitewing in the same day for 15 minutes.
  All of the bitewing radiographs will be evaluated by two experienced restorative dentists for caries. All observers will be instructed on the definition of the rating scale before the examination sessions. The observers will be using the following a 5-point confidence scale as follows: 1=caries definitely absent; 2=caries probably absent; 3=equal chance of caries being present or absent; 4=caries probably present; 5=caries definitely present. If caries was detected a second 5-point confidence scale as follows: 1=caries mostly absent (< 25%); 2=caries slightly presence( 25%-50%) ; 3=about half of the border are presence; 4=caries probably clear ( most boarders are presence); 5=caries definitely clear ( all borders are presence ).
- Horizontal Bitewing, Then Vertical Bitewing: Participants first received horizontal bitewing in one day for 15 minutes . After a washout period of 10 minutes, they then received vertical bitewing in the same day for 15 minutes.
  All of the bitewing radiographs will be evaluated by two experienced periodontist for bone loss measurements. The steel wire will be used to determine the magnification factor as explained by G Li et al. 8 The steel wire and cemento enamel junction (CEJ) - if not obscure by caries - will be used as reference points for bone loss measurements. Each tooth will be measured mesially and distally twice and all these measurements will be adjusted using the steel measurement.9 All the measurements will be conducted using IC measure INK software.
Period: First Intervention (15 Minutes)
Arm/Group | Vertical Bitewing, Then Horizontal Bitewing | Horizontal Bitewing, Then Vertical Bitewing
Started | 10 | 10
Completed (This is a cross over study design .So, we have 20 patients but they act as a case and control .So, they look like 40 .) | 10 | 10
Not Completed | 0 | 0
Period: Washout (10 Minutes)
Arm/Group | Vertical Bitewing, Then Horizontal Bitewing | Horizontal Bitewing, Then Vertical Bitewing
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention (15 Minutes)
Arm/Group | Vertical Bitewing, Then Horizontal Bitewing | Horizontal Bitewing, Then Vertical Bitewing
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Vertical Bitewing, Then Horizontal Bitewing: Participants first received vertical bitewing. After a washout period of 15 min, they then received Horizontal bitewing.
- Experimental: Horizontal Bitewing, Then Vertical Bitewing: Participants first received horizontal bitewing. After a washout period of 15 min, they then received vertical bitewing.
- Total: Total of all reporting groups
Arm/Group | Experimental: Vertical Bitewing, Then Horizontal Bitewing | Experimental: Horizontal Bitewing, Then Vertical Bitewing | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.05 (9.79) | 25.74 (12.83) | 29.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 4 | 2 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of radiography [Mean (Standard Deviation); unit: x ray] | 5.9 (1.7) | 5.3 (1.3) | 5.6 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Caries Detection
Description: Count number of teeth with caries
Time Frame: baseline and 15 minutes
Measure: Mean (95% Confidence Interval); unit: teeth
Units Other Than Participants: Teeth
Groups:
- Vertical Bitewing: Participants who received vertical bitewing in either the first or last 15 minutes of the study.
- Horizontal Bitewing: Participants who received horizontal bitewing in either the first or last 15 minutes of the study.
Arm/Group | Vertical Bitewing | Horizontal Bitewing
Number analyzed (Participants) | 10 | 10
Number analyzed (Teeth) | 320 | 320
teeth | 7.22 [6.00 to 8.44] | 6.48 [5.24 to 7.72]

2. Primary Outcome: Level of Bone Loss
Description: All of the bitewing radiographs will be evaluated for bone loss measurements. The steel wire will be used to determine the magnification factor . The steel wire and cemento enamel junction (CEJ) - if not obscure by caries - will be used as reference points for bone loss measurements. Each tooth will be measured from the CEJ to the bone crest.
Time Frame: baseline and at 15 minutes
Measure: Mean (Standard Deviation); unit: mm of bone loss
Units Other Than Participants: Teeth
Arm/Group | Vertical Bitewing | Horizontal Bitewing
Number analyzed (Participants) | 20 | 20
Number analyzed (Teeth) | 320 | 320
mm of bone loss | 1.15 (0.69) | 1.12 (0.63)

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Vertical Bitewing: Participants first received vertical bitewing in one day for 15 minutes . After a washout period of 10 minutes, they then received horizontal bitewing in the same day for 15 minutes.
- Horizontal Bitewing: Participants first received horizontal bitewing in one day for 15 minutes . After a washout period of 10 minutes, they then received vertical bitewing in the same day for 15 minutes.
Arm/Group | Vertical Bitewing | Horizontal Bitewing
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT04341636/Prot_SAP_000.pdf